CLINICAL TRIAL: NCT06870448
Title: Methylprednisolone With Endovascular Thrombectomy for Large Ischemic Stroke (MATCH): A Randomized Controlled Trial
Brief Title: Methylprednisolone With Endovascular Thrombectomy for Large Ischemic Stroke
Acronym: MATCH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYS-5010-202501
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: large infarct core; methylprednisolone; endovascular thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone group (Experimental): Methylprednisolone sodium succinate
  Interventions: Drug: Methyprednisolone sodium succinate
- Placebo group (Placebo Comparator): Methylprednisolone sodium succinate simulant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methyprednisolone sodium succinate — Methylprednisolone at a dose of 2 mg/kg/day for 3 consecutive days, with a maximum daily dose of 160 mg (4 vials, 40 mg per vial, Hanhui Pharmaceutical Co., Ltd.). The initial study drug will be administered as soon as possible after randomization. It is recommended that the initial study drug be administered before arterial access closure.
  Other Names: Methylprednisolone
  Arms: Methylprednisolone group
Drug: Placebo — Placebo for 3 consecutive days, with a maximum daily dose of 4 vials (Hanhui Pharmaceutical Co., Ltd.)
  Other Names: Methylprednisolone sodium succinate simulant
  Arms: Placebo group

SUMMARY:
It is uncertain whether intravenous methylprednisolone improves outcomes for acute anterior circulation large vascular occlusion (LVO) patients with a large infarct core. In this study, the investigators assume that methylprednisolone plus endovascular thrombectomy (EVT) might be superior to EVT alone for patients who have evidence of a large infarct volume. The objective of the study was to establish the efficacy and safety of methylprednisolone with EVT in patients presenting with symptoms of acute ischemic stroke from LVO in the anterior circulation and having a large infarct volume.

DETAILED DESCRIPTION:
MATCH is a multicentered, prospective, randomized, controlled trial. A total of 1614 patients (age ≥18 years) with NIHSS ≥6 and pre-stroke modified Rankin Scale (mRS) 0-2, within 24 hours of symptom onset of acute ischemic stroke, who has the imaging evidence of an occlusion of the intracranial internal carotid artery (ICA) and/or M1/M2 segment of middle cerebral artery (MCA), large infarct core [defined as: 1) NCCT (non-contrast computed tomography) ASPECTS (Alberta Stroke Program Early CT Score) 0-5, decided on last head CT scan before randomization. Or 2) Ischemic core volume ≥70ml, determined either on a diffusion-weighted MRI map based on an ADC (Apparent Diffusion Coefficient) threshold of less than 620 or on CTP (computed tomography perfusion) image with rCBF<30%] will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content. One group will receive methylprednisolone plus EVT, the other group will receive methylprednisolone simulant plus EVT. The primary objective is to evaluate the efficacy of methylprednisolone with EVT in patients presenting with symptoms of acute ischemic stroke from LVO in the anterior circulation and having a large infarct volume. The study consists of four visits including the day of randomization, 36 hours after randomization, 7 days or discharge, and 90 days. The primary outcome is a shift in the distribution of scores on the mRS at 90 days. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee (EC) in Sun Yat-Sen Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years;
* 2. Clinically diagnosed with acute ischemic stroke and NIHSS ≥6;
* 3. CT angiography (CTA), MR angiography (MRA) or digital subtraction angiography (DSA) confirmed occlusion of intracranial internal carotid artery (ICA) or M1/M2 segments of middle cerebral artery (MCA) and plan to undergo EVT;
* 4. ASPECTS ≤5 (based on NCCT) or infarct core volume ≥70mL (defined as rCBF <30% on CT perfusion or ADC <620 on MRI);
* 5. Time from symptom onset to randomization within 24 hours (from last known well);
* 6. Pre-stroke mRS score 0-2;
* 7. Written informed consent signed by patients or their family members.

Exclusion Criteria:

* 1. Intracranial hemorrhage confirmed by CT or MRI;
* 2. Allergic to glucocorticoids or placebo components;
* 3. Allergic to contrast agent;
* 4. Presence of severe infectious disease unsuitable for glucocorticoid therapy or any other contraindication to glucocorticoid use;
* 5. Known genetic or acquired coagulopathy, coagulation factor deficiency, use of warfarin with an international normalized ratio (INR) >1.7, or use of novel oral anticoagulants within 48 hours of symptom onset;
* 6. Platelet count <90×10^9/L;
* 7. Random blood glucose <2.8 mmol/L or >22.2 mmol/L;
* 8. History of gastrointestinal or urinary tract bleeding within the last month;
* 9. Current participation in another interventional clinical study;
* 10. Pregnant or lactating women;
* 11. Renal dysfunction (glomerular filtration rate <30 ml/min or serum creatinine >220 μmol/L [2.5 mg/dl]);
* 12. Uncontrolled hypertension with persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, refractory to medical management;
* 13. Life expectancy less than 6 months due to malignancy or severe cardiopulmonary disease;
* 14. Other conditions deemed unsuitable for the study by the investigator, such as inability to comprehend or comply with study procedures or follow-up due to mental illness, cognitive or emotional disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1614 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
90-day distribution of patients across the ordinal modified Rankin Scale (mRS) | 90±14 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms. Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) 0-1 at 90±14 days | 90±14 days after randomization
  Excellent functional outcome defined as a modified Rankin Scale (mRS) score of 0-1 at 90±14 days
modified Rankin Scale (mRS) 0-2 at 90±14 days | 90±14 days after randomization
  Good clinical outcome defined as a modified Rankin Scale (mRS) score of 0-2 at 90±14 days
modified Rankin Scale (mRS) 0-3 at 90±14 days | 90±14 days after randomization
  Independent ambulation defined as a modified Rankin Scale (mRS) score of 0-3 at 90±14 days
modified Rankin Scale (mRS) 0-4 at 90±14 days | 90±14 days after randomization
  No constant care required defined as modified Rankin Scale (mRS) 0-4 at 90±14 days
Quality of Life (EuroQoL 5-Dimension 5-Level) at 90±14 days | 90±14 days after randomization
  The value of Quality of Life (EuroQoL 5-Dimension 5-Level) at 90±14 days
National Institutes of Health Stroke Scale (NIHSS) score change from baseline | 7±1 days after randomization/discharge
  National Institutes of Health Stroke Scale (NIHSS) score change from baseline, at 7 (±1) days or at discharge
Infarct core volume change from baseline | 7±1 days after randomization/discharge or at 36±12 hours after randomization
  Infarct core volume change from baseline, assessed with NCCT at 7±1 days after randomization/at discharge or with MRI at 36±12 hours
Rate of hemicraniectomy within 7 days | 7±1 days after randomization/discharge
  Rate of hemicraniectomy

OTHER OUTCOMES:
All-cause mortality within 90 days (Safety Outcome) | 90±14 days after randomization
  All-cause mortality within 90 days
Time to all-cause mortality within 90 days (Safety Outcome) | Randomization up to 90±14 days after randomization
  Time to all-cause death is defined as the time from randomization to the time of death
Rate of symptomatic intracranial hemorrhage (sICH) per Heidelberg Bleeding Classification within 48 hours (Safety Outcome) | 36±12 hours after randomization
  Heidelberg Bleeding Classification was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below:
  * 4 points total NIHSS at the time of diagnosis compared to immediately before worsening.
  * 2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention.
  Absence of alternative explanation for deterioration.
Any serious adverse events and steroid-related adverse events (hyperglycemia, infection, gastrointestinal hemorrhage) within 90 days (Safety Outcome) | From the signing of informed consent up to 90±14 days after randomization
  Safety will be assessed according to common terminology criteria for adverse events version 5.0 (CTCAE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Qingyu Shen, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from principal investigator upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion
Access Criteria: The IPD will be available from principal investigator upon reasonable request.